CLINICAL TRIAL: NCT06685731
Title: The Effects of Laughter Yoga on Sleep Quality, Vitality, Active Aging, and Quality of Life in Elderly Individuals
Brief Title: Laughter Yoga is Role in Enhancing Sleep and Well-being in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Şerife Köleoğlu, Lecturer, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Artvin Çoruh Universty
Record Dates: First submitted 2024-09-05; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: ELDERLY PEOPLE
Keywords: elderly; Laughter Yoga; Sleep Quality; Vitality; Active Aging; Elderly Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group (Experimental): Personal Information Form, Mini-Mental State Examination, Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for Elderly Individuals will be administered to elderly individuals via face-to-face interviews conducted by the researcher.
  Elderly individuals will be provided with information about the Laughter Yoga sessions.
  The elderly participants will undergo a total of 12 Laughter Yoga sessions, with each session lasting 40 minutes, conducted twice a week for 6 weeks.
  Participants' phone numbers will be collected, and they will be contacted twice a week to ensure their attendance at the Laughter Yoga sessions.
  Interventions: Other: Laughter Yoga
- Control group (No Intervention): Personal Information Form, Mini-Mental State Examination, Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly will be administered to elderly individuals through face-to-face interviews conducted by the researcher.
  No intervention will be applied to the elderly individuals in this group.
  Phone numbers of the participants in this group will be collected, and they will be contacted once a week to check on their status.

INTERVENTIONS:
Other: Laughter Yoga — Laughter Yoga Intervention:
  Laughter Yoga is composed of four stages: deep breathing exercises, clapping and warm-up exercises, childlike play, and laughter exercises. These stages are designed to remove barriers to laughter, enhance emotional expression through childlike play, and prepare the lungs for laughter exercises.
  Before the Laughter Yoga session begins, participants will be introduced to both the practice itself and to Laughter Yoga in general. The session will then proceed according to the following structure:
  Deep Breathing Exercises: Participants inhale through the nose for 4-5 seconds, hold their breath for 2-3 seconds, and exhale through the mouth, with lips pursed, for one second longer than the inhalation, while smiling or laughing. This exercise is performed for 10-15 minutes.
  Clapping and Warm-Up Exercises: Participants clap with palms and fingertips touching, keeping their hands parallel. This stimulates acupressure points in the hands. To increase group energy, a
  Other Names: Laughter Therapy
  Arms: Participant Group

SUMMARY:
Objective:

The study aims to evaluate the effects of Laughter Yoga on sleep quality, vitality, active aging, and quality of life in individuals aged 60 and over.

Method:

This randomized controlled experimental study will be conducted between 01.09.2024 and 31.12.2024 with elderly individuals aged 60 and over who are registered at Şavşat Family Health Center No. 1. The study population consists of 6,797 individuals. Participants will be randomly assigned to an experimental group (30) and a control group (30) using a simple randomization method. Data will be collected using a Personal Information Form, Mini-Mental State Examination, Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly. The experimental group will participate in 12 Laughter Yoga sessions, conducted twice a week for 6 weeks, with each session lasting 40 minutes. No intervention will be applied to the control group. At the end of the 6th week, final measurements will be taken from both groups at the family health center.

DETAILED DESCRIPTION:
Laughter yoga offers various approaches and insights related to humor, is low-cost, and can be easily practiced regardless of time and place, making it a highly effective and practical intervention. Research on the physiological health effects of laughter yoga has demonstrated that it enhances muscle activation, relaxes muscles, increases respiratory rate, stimulates circulation, improves oxygen saturation, reduces stress hormones (e.g., adrenaline, noradrenaline, cortisol), elevates beta-endorphin levels, alleviates pain, and enhances cognitive function. Additionally, the positive effects of humor and emotions such as happiness and optimism on psychosocial health are well-recognized. Studies on the psychosocial health outcomes of laughter yoga indicate that it reduces stress, anxiety, and depression, while improving mood, self-esteem, self-efficacy, happiness, optimism, and energy levels. Furthermore, it helps reduce interpersonal conflicts and tensions, enhances social relationships and quality of life, and boosts psychological well-being.

Although the use of laughter yoga among older adults is limited, research has shown that it has a positive impact on depression, anxiety, sleep quality, quality of life, loneliness, life satisfaction, blood pressure, and pain in this population.A review of the literature suggests that laughter yoga may be effective in improving certain physiological and psychosocial health outcomes, highlighting the need for further research.

This study aims to evaluate the effectiveness of laughter yoga in nursing practice, support its application, and investigate its potential benefits for elderly individuals. Specifically, it seeks to assess its positive impact on sleep quality, vitality, active aging, and overall quality of life, while confirming that it poses no adverse side effects for older adults.

Elderly individuals registered at the family health center will be introduced to the study and provided with detailed information regarding its objectives. Those who meet the inclusion criteria and express interest in participating will be identified. After obtaining informed consent, participants will be assigned to groups according to a randomization list. The researcher has obtained an "International Laughter Yoga Leadership Certificate" to conduct the Laughter Yoga intervention within the scope of this study.

The Personal Information Form, Mini-Mental State Examination, Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly will be administered to both groups through face-to-face interviews conducted by the researcher (pre-test). Participants in the experimental group will be provided with comprehensive information about the Laughter Yoga intervention.

The experimental group will participate in 12 Laughter Yoga sessions, conducted twice a week over a 6-week period, with each session lasting 40 minutes. As the contagious nature of laughter facilitates easier participation when group size is larger, participants will not be divided into smaller groups during the Laughter Yoga sessions. The sessions will be led by the researcher, and their duration and frequency have been determined based on a thorough review of the relevant literature. Sessions will be held in the gymnasium of the institution where the researcher is employed, under optimal conditions. No intervention will be applied to the control group. At the end of the 6th week, participants from both groups will be invited to the family health center, where the Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly will be administered again (post-test).

Participants in both groups will continue using their routine medications throughout the 6-week study period. Upon completion of the research, elderly individuals in the control group will be offered information on Laughter Yoga upon request.

Elderly individuals registered at the family health center will be introduced to the study and provided with detailed information regarding its objectives. Those who meet the inclusion criteria and express interest in participating will be identified. After obtaining informed consent, participants will be assigned to groups according to a randomization list. The researcher has obtained an International Laughter Yoga Leadership Certificate to conduct the Laughter Yoga intervention within the scope of this study.

The Personal Information Form, Mini-Mental State Examination, Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly will be administered to both groups through face-to-face interviews conducted by the researcher (pre-test). Participants in the experimental group will be provided with comprehensive information about the Laughter Yoga intervention.

The experimental group will participate in 12 Laughter Yoga sessions, conducted twice a week over a 6-week period, with each session lasting 40 minutes. As the contagious nature of laughter facilitates easier participation when group size is larger, participants will not be divided into smaller groups during the Laughter Yoga sessions. The sessions will be led by the researcher, and their duration and frequency have been determined based on a thorough review of the relevant literature. Sessions will be held in the gymnasium of the institution where the researcher is employed, under optimal conditions. No intervention will be applied to the control group. At the end of the 6th week, participants from both groups will be invited to the family health center, where the Active Aging Scale, Pittsburgh Sleep Quality Index, Subjective Vitality Scale, and Quality of Life Scale for the Elderly will be administered again (post-test).

Participants in both groups will continue using their routine medications throughout the 6-week study period. Upon completion of the research, elderly individuals in the control group will be offered information on Laughter Yoga upon request.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Şavşat,
* Aged 60 or over,
* No issues with vision, hearing, or perception,
* Scored 24 or higher on the Mini-Mental State Examination,
* Not undergoing psychiatric treatment,
* No physical limitations that would impede participation in laughter yoga (e.g., fractures, open wounds, or muscle weakness in the hands, wrists, or arms),
* Literate,
* Open to communication,
* Willing to participate in the study.

Exclusion Criteria:

* Scored below 24 on the Mini-Mental State Examination,
* Severe hearing or perceptual impairments that hinder communication,
* Major psychiatric disorders,
* Underwent surgery within the last three months,
* Medical conditions that could cause physical strain or increase abdominal pressure during laughter yoga (e.g., bleeding hemorrhoids, any type of hernia, persistent cough, severe back pain, heart disease, hypertension, urinary incontinence, epilepsy), and individuals with oncological conditions will be excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-test | Initial enrollment in the study
  Mini Mental State Test (MMST): Assesses cognitive function on a 0-30 scale; higher scores indicate better cognitive function. The score will be reported independently.

SECONDARY OUTCOMES:
Active Aging Scale | From enrollment to the end of treatment at 6 weeks
  Scores range from 0 to 272 across four subscales, with higher scores indicating greater active aging. This score is reported as a separate outcome.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 6 weeks
  Measures sleep quality, where scores of 5 or more indicate poor sleep quality. PSQI results are reported separately.
Subjective Vitality Scale (SVS) | From enrollment to the end of treatment at 6 weeks
  Ranges from 7 to 49, with higher scores reflecting higher vitality. It is reported as an independent measure of vitality.
CASP-13 Quality of Life Scale | From enrollment to the end of treatment at 6 weeks
  Evaluates quality of life in terms of autonomy and satisfaction, with higher scores indicating better life quality, and will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Tan, Prof. Dr., Study Director — Atatürk Universty
Locations (1):
- Şavşat 1St Family Health Center, Artvin, Şavşat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No